CLINICAL TRIAL: NCT03717974
Title: Randomized Controlled Pilot Study for Medico-economic Impact Evaluation in Telemedecine Follow-up in Complement of a Mobile Team in Patients With Neurological Disabilities (HANDI@CCESS)
Brief Title: Medico-economic Impact Evaluation in Telemedecine Follow-up in Complement of a Mobile Team in Patients With Neurological Disabilities (HANDI@CCESS)
Acronym: HANDI@CCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Collaborators: Clinique Mutualiste la Sagesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-A02378-45
Record Dates: First submitted 2018-10-16; First posted 2018-10-24 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2021-02

CONDITIONS: Severe Neurological Disabilities
Keywords: telemedecine; medico-economic; neurological disability

STUDY DESIGN:
Intervention Model Description: Monocentric, randomized controlled pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telemedecine's follow-up (Experimental): Telemedecine follow-up after an intervention at home of the mobile team
  Interventions: Other: Telemedecine follow-up after an intervention at home of the mobile team
- mobile team's follow-up (Active Comparator): Mobile team follow-up after an intervention at home of the mobile team
  Interventions: Other: Mobile team follow-up after an intervention at home of the mobile team

INTERVENTIONS:
Other: Telemedecine follow-up after an intervention at home of the mobile team — After a first visit of the mobile team at home, patients are followed by telemedicine. Moreover, in case of pain, a specialized consultation by an algologist of "La Sagesse" will be realized.
  Other Names: medico-economic analysis
  Arms: telemedecine's follow-up
Other: Mobile team follow-up after an intervention at home of the mobile team — After a first visit of the mobile team at home, patients are followed by mobile team. Moreover, in case of pain, a specialized consultation by an algologist of "La Sagesse" will be realized.
  Other Names: medico-economic analysis
  Arms: mobile team's follow-up

SUMMARY:
Access to care for people with traumatic or degenerative neurological disabilities is a current public health concern. New technological tools such as telemedicine can bring expertise to the place of life of people while promoting the city-hospital link.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18
* Volunteer to participate in the study and whose primary caregiver is voluntary
* Presenting a severe neurological handicap following a neurological lesion of traumatic, vascular or degenerative origin,
* Requiring an expert opinion in MPR (rehabilitation, technical and human compensatory means, specific treatments ...) and / or in algology
* Whose access to care is reduced (difficulties of movement, distance from expert centers, situation of fragility ...) and which necessitate the displacement of professionals at home,
* Which require a coordination of care associating the professionals of the sanitary and medico-social sectors
* Living in health territory 5 in Brittany
* Mastering the French language spoken and / or written.

Exclusion Criteria:

* Misunderstanding making it impossible for informed consent with the refusal of the guardian or court safeguard
* Unable to use a digital tablet or lack of a resource person who can assist the patient in the use of the tablet
* Patients who do not have access to an internet connection (white area)
* Life threatening is committed in the short term (< 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Medical-economic analysis by the calculation of the cost-effectiveness of this organization of care | 6 months
  Cost-effectiveness analysis by ICER (Incremental Cost-Effectiveness Ratio)

SECONDARY OUTCOMES:
UTAUT (Unified theory of acceptance of technology) questionnaire | 6 months
  Questionnaire of acceptability / acceptance of the tool and its use by professionals based on the Unified Theory of Acceptance and Use Technology (UTAUT)
Hospital Anxiety and Depression scale (HAD) | 6 months
  It can detect anxiety and depressive disorders. It has 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus obtaining two scores (maximum score of each score = 21). 7 or less: no symptomatology 8 to 10: doubtful symptomatology 11 and above: certain symptomatology.
Pain evaluation | 6 months
  Digital assessment (0 to 10) of pain for communicating patients
DN4 scale | 6 months
  Digital assessment of neuropathic pain for communicating patients. If the patient score is equal to or greater than 4/10, the test is positive.
Doloplus scale | 6 months
  Behavioral Assessment Scale of Pain in Older People with Verbal Communication Disorders. This scale comprises ten items divided into three subgroups (five somatic, two psychomotor and three psychosocial).
  Each item is rated from 0 to 3 (four exclusive and progressive level scoring), which results in an overall score between 0 and 30.
  The pain is clearly affirmed for a score greater than or equal to 5 out of 30.
Zarit's score | 6 months
  The Zarit scale assesses the emotional, physical and financial burden for caregivers of caring for someone with a loss of autonomy.
  The total score, which is the sum of the scores obtained for each of 22 items, varies from 0 to 88.
  A score less than or equal to 20 indicates a low or no load; a score between 21 and 40 indicates a light load; a score between 41 and 60 indicates a moderate load; a score above 60 indicates a severe charge.
Goal Attainment Scale | 6 months
  Goal Attainment Scale by objectives at the beginning and end of taking charge. Each item built has 5 levels of answers 0: corresponds to the achievement of the goal set by the examiner.
  * 1: is a better score than expected.
  * 2: corresponds to the most favorable evolution expected.
    * 1: corresponds to a score lower than that expected.
    * 2: corresponds to a least favorable score expected.
EVA Satisfaction | 6 months
  Digital assessment (0 to 10) of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gallien, Doctor, Principal Investigator — Pole Saint-Hélier
Locations (1):
- Pôle Saint-Hélier, Rennes, France

IPD SHARING:
Plan to Share IPD: No